CLINICAL TRIAL: NCT02572752
Title: Bioequivalence of 1 Soft Gelatine Capsule Containing 200 mg Nintedanib Compared to 2 Soft Gelatine Capsules Containing 100 mg Nintedanib Following Oral Administration in Healthy Male Subjects
Brief Title: Relative Bioavailability of 2 Oral Formulations of Nintedanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199.237; 2015-001348-12 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib

ARMS (3):
- Treatment T (Test) (Experimental): Nintedanib, 1 capsule, oral with 240 mL of water
  Interventions: Drug: Nintedanib
- Treatment R - 1 (Reference) (Experimental): Nintedanib, 2 capsules, oral with 240 mL of water
  Interventions: Drug: Nintedanib
- Treatment R - 2 (Reference) (Experimental): Nintedanib, 2 capsules, oral with 240 mL of water
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — 1 soft gelatine capsule, single dose, oral
  Arms: Treatment T (Test)
Drug: Nintedanib — Nintedanib, 2 soft gelatine capsules, single dose, oral
  Arms: Treatment R - 1 (Reference)
Drug: Nintedanib
  Other Names: Nintedanib, 2 soft gelatine capsules, single dose, oral
  Arms: Treatment R - 2 (Reference)

SUMMARY:
To establish the bioequivalence of 1 soft gelatine capsule containing 200 mg nintedanib compared to 2 soft gelatine capsules containing 100 mg nintedanib

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests.
2. Age of 18 to 50 years (incl.)
3. Body weight of at least 70 kg
4. BMI of 21 to 31 kg/m2 (incl.)
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
6. Male subjects, who are willing to use a medically acceptable method of contraception during the first 3 months after administration of nintedanib. Acceptable methods of contraception for use by male volunteers include sexual abstinence, a vasectomy performed at least 1 year prior to dosing and barrier contraception (condom). Subjects, who are not vasectomised or sexually abstinent have to ensure that an additional acceptable method of contraception will be used by his female partner such as IUD (intrauterine device), surgical sterilisation (including hysterectomy), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first nintedanib administration, or barrier method (e.g. diaphragm with spermicide).

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts
9. Chronic or relevant acute infections
10. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
11. Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
12. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
13. Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
14. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
15. Inability to refrain from smoking on specified trial days
16. Alcohol abuse (consumption of more than 30 g per day for males)
17. Drug abuse or positive drug screening
18. Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
19. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
20. Inability to comply with dietary regimen of trial site
21. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was randomised and open-label with a 3-way crossover design (2 administrations of reference treatment and 1 administration of test treatment in all subjects). In this study 70 subjects were entered and treated.
Groups:
- Nin 2x100 mg(R1) / Nin 2x100 mg(R2) / Nin 1x200 mg(T): Subjects were treated with single oral dose, started in Period 1 (Reference treatment (R1)) and Period 2 (Reference treatment (R2)) with nintedanib (nin) soft gelatine capsule, 200 mg (2x100 mg) with about 240 mL of water, followed in Period 3 (Test treatment (T)) with nintedanib soft gelatine capsule, 200 mg (1x200mg) with about 240 mL of water. Treatment periods were separated by a wash-out phase of at least 12 days.
- Nin 2x100 mg(R1) / Nin 1x200 mg(T) / Nin 2x100 mg(R2): Subjects were treated with single oral dose, started in Period 1 (Reference treatment (R1)) with nintedanib soft gelatine capsule, 200 mg (2x100mg) with about 240 mL of water, followed in Period 2 (Test treatment (T)) with nintedanib soft gelatine capsule, 200 mg (1x200mg) with about 240 mL of water and in Period 3 (Reference treatment (R2)) with nintedanib soft gelatine capsule, 200 mg (2x100mg) with about 240 mL of water. Treatment periods were separated by a wash-out phase of at least 12 days.
- Nin 1x200 mg(T) / Nin 2x100 mg(R1) / Nin 2x100 mg(R2): Subjects were treated with single oral dose, started in Period 1 (Test treatment (T)) with nintedanib soft gelatine capsule, 200 mg (1x200mg) with about 240 mL of water, followed in Period 2 (Reference treatment (R1)) and Period 3 (Reference treatment (R2)) with nintedanib soft gelatine capsule, 200 mg (2x100 mg) with about 240 mL of water. Treatment periods were separated by a wash-out phase of at least 12 days.
Period: Period 1 Including Washout
Arm/Group | Nin 2x100 mg(R1) / Nin 2x100 mg(R2) / Nin 1x200 mg(T) | Nin 2x100 mg(R1) / Nin 1x200 mg(T) / Nin 2x100 mg(R2) | Nin 1x200 mg(T) / Nin 2x100 mg(R1) / Nin 2x100 mg(R2)
Started | 23 | 23 | 24
Completed | 23 | 23 | 24
Not Completed | 0 | 0 | 0
Period: Period 2 Including Washout
Arm/Group | Nin 2x100 mg(R1) / Nin 2x100 mg(R2) / Nin 1x200 mg(T) | Nin 2x100 mg(R1) / Nin 1x200 mg(T) / Nin 2x100 mg(R2) | Nin 1x200 mg(T) / Nin 2x100 mg(R1) / Nin 2x100 mg(R2)
Started | 23 | 23 | 24
Completed | 23 | 23 | 24
Not Completed | 0 | 0 | 0
Period: Period 3 Including Washout
Arm/Group | Nin 2x100 mg(R1) / Nin 2x100 mg(R2) / Nin 1x200 mg(T) | Nin 2x100 mg(R1) / Nin 1x200 mg(T) / Nin 2x100 mg(R2) | Nin 1x200 mg(T) / Nin 2x100 mg(R1) / Nin 2x100 mg(R2)
Started | 23 | 23 | 24
Completed | 23 | 23 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This analysis set included all 70 subjects (that is, all subjects who received at least 1 dose of study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | Nin 2x100 mg(R1) / Nin 2x100 mg(R2) / Nin 1x200 mg(T) | Nin 2x100 mg(R1) / Nin 1x200 mg(T) / Nin 2x100 mg(R2) | Nin 1x200 mg(T) / Nin 2x100 mg(R1) / Nin 2x100 mg(R2) | Total
Number analyzed (Participants) | 23 | 23 | 24 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (10.3) | 36.6 (9.5) | 31.6 (7.2) | 34.0 (9.2)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 23 | 23 | 24 | 70

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). The unadjusted geometric mean (gMean) and geometric coefficient variation (gCV) was calculated for Test treatment (T), Reference treatment 1 (R1) and Reference treatment 2 (R2) separately.
Time Frame: -1:00 hour(h) before drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 3:30h, 4:00h, 4:30h, 5:00h, 5:30h, 6:00h, 7:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h and 72:00h after drug administration.
Population: Pharmacokinetic Set (PKS) : This analysis set included all treated subjects who provided at least 1 observation for at least 1 primary endpoint, and who had no important protocol violations impacting statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Nintedanib, Test Treatment (T): Subjects were treated with single oral dose, started in Period 1 (Test treatment (T)) with nintedanib soft gelatine capsule, 200 mg (1x200mg) with about 240 mL of water.
- Nintedanib, Reference Treatment (R1): Subjects were treated with single oral dose, started in Period 1 (Reference treatment (R1)) with nintedanib soft gelatine capsule, 200 mg (2x100mg) with about 240 mL of water.
- Nintedanib, Reference Treatment (R2): Subjects were treated with single oral dose, started in Period 1 (Reference treatment (R2)) with nintedanib soft gelatine capsule, 200 mg (2x100mg) with about 240 mL of water.
Arm/Group | Nintedanib, Test Treatment (T) | Nintedanib, Reference Treatment (R1) | Nintedanib, Reference Treatment (R2)
Number analyzed (Participants) | 70 | 70 | 70
ng*h/mL | 300 (38.8) | 310 (37.6) | 306 (36.2)
Statistical Analysis 1: Comparison: Nintedanib, Test Treatment (T) vs Nintedanib, Reference Treatment (R1) vs Nintedanib, Reference Treatment (R2); An Analysis of variance (ANOVA) model was used on the logarithmic scale in order to compare the Test treatment vs. the Reference treatment (without differentiation between R1 and R2). This model included effects for 'sequence', 'subjects within sequences', 'period' and 'treatment'. For the two 1-sided t-test procedure, the effect 'subjects within sequences' was considered to be random, whereas the other effects were considered to be fixed; Test type: Superiority or Other; p < 0.0001, ANOVA; gMean Ratio = 97.478, 90% CI 2-sided [94.545 to 100.502], Standard Error of Mean 11.57 — Relative bioavailability was estimated by the ratios of the gMean of nin Test treatment (T) divided by nin Reference treatment (R1 & R2). Standard Error of the mean is actually the intra individual geometric coefficient variation (gCV)

2. Primary Outcome: Cmax
Description: Maximum measured concentration of the analyte in plasma (Cmax). The unadjusted geometric mean (gMean) and geometric coefficient variation (gCV) was calculated for Test treatment (T), Reference 1 treatment (R1) and Reference 2 treatment (R2) separately.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib, Test Treatment (T) | Nintedanib, Reference Treatment (R1) | Nintedanib, Reference Treatment (R2)
Number analyzed (Participants) | 70 | 70 | 70
ng/mL | 39.3 (56.0) | 41.1 (43.4) | 39.8 (46.3)
Statistical Analysis 1: Comparison: Nintedanib, Test Treatment (T) vs Nintedanib, Reference Treatment (R1) vs Nintedanib, Reference Treatment (R2); An ANOVA model was used on the logarithmic scale in order to compare the Test treatment vs. the Reference treatment (without differentiation between R1 and R2). This model included effects for 'sequence', 'subjects within sequences', 'period' and 'treatment'. For the two 1-sided t-test procedure, the effect 'subjects within sequences' was considered to be random, whereas the other effects were considered to be fixed; Test type: Superiority or Other; p < 0.0001, ANOVA; gMean Ratio = 97.004, 90% CI 2-sided [90.948 to 103.463], Standard Error of Mean 20.77 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC0-inf
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf). The unadjusted geometric mean (gMean) and geometric coefficient variation (gCV) was calculated for Test treatment (T), Reference 1 treatment (R1) and Reference 2 treatment (R2) separately.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib, Test Treatment (T) | Nintedanib, Reference Treatment (R1) | Nintedanib, Reference Treatment (R2)
Number analyzed (Participants) | 70 | 70 | 70
ng*h/mL | 311 (38.8) | 322 (37.7) | 319 (36.4)
Statistical Analysis 1: Comparison: Nintedanib, Test Treatment (T) vs Nintedanib, Reference Treatment (R1) vs Nintedanib, Reference Treatment (R2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; gMean Ratio = 97.149, 90% CI 2-sided [94.223 to 100.166], Standard Deviation 11.40 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 12 days after the last drug administration of nintedanib, ie., upto 16 days.
Groups:
- Nintedanib, Test Treatment (T): Subjects were treated with single oral dose of nintedanib soft gelatine capsule (Test treatment (T)) , 200 mg (1x200mg) with about 240 mL of water.
- Nintedanib, Reference Treatment (R1 & R2): Subjects were treated twice with single oral dose of nintedanib soft gelatine capsule (Reference treatment (R1 & R2)), 200 mg (2x100mg) with about 240 mL of water.
Arm/Group | Nintedanib, Test Treatment (T) | Nintedanib, Reference Treatment (R1 & R2)
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 24/70 | 29/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib, Test Treatment (T) (N=70) | Nintedanib, Reference Treatment (R1 & R2) (N=70)
Diarrhoea (Gastrointestinal disorders) | 16 | 20
Nausea (Gastrointestinal disorders) | 4 | 6
Nasopharyngitis (Infections and infestations) | 2 | 4
Headache (Nervous system disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes